CLINICAL TRIAL: NCT02072772
Title: A Trial of Positively Smoke Free Group Therapy for HIV-infected Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Georgetown University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-260; R01DA036445-01 (NIH)
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Tobacco Use in Persons Living With HIV
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positively Smoke Free group treatment (Experimental): Eight 90 minute group sessions (6-8 HIV-infected smokers per group) led by a pair of trained group leaders: a "professional" with psychology or social work training and a "peer" HIV-infected ex-smoker with tobacco treatment training.
  All subjects will be offered a 3 month supply of nicotine patches
  Interventions: Behavioral: Positively Smoke Free group treatment
- Standard care (Active Comparator): Brief (<5 minutes) advice to quit Offer of nicotine patches Self-help brochure
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Positively Smoke Free group treatment — See Arm Description
  Arms: Positively Smoke Free group treatment
Behavioral: Standard Care — See Arm Description
  Arms: Standard care

SUMMARY:
The purpose of this study is to determine whether Positively Smoke Free group therapy is more effective at promoting cessation than standard care.

DETAILED DESCRIPTION:
There are 1.1 million persons living with HIV (PLWH) in the US, 60% of them smoke cigarettes, and 75% of these are interested in quitting. Almost none are currently accessing smoking cessation interventions designed to meet their specific needs and concerns.

Cigarette smoking is responsible for 24% of deaths among PLWH, and 30% of non-AIDS defining malignancies. It is driving the alarming rise in cardiac events and lung cancers in this highly vulnerable population. The lack of access to proven, effective, culturally appropriate tobacco cessation services represents a health disparity of the first order. The psychosocial profile of the PLWH-smoker community, characterized by high rates of psychiatric comorbidity, drug and alcohol use, and low levels of social support, suggests that achieving high cessation rates will be a great challenge.

Positively Smoke Free (PSF) is an intensive, multisession, group cessation program specifically developed for PLWH smokers. A pilot study of PSF yielded promising results. This proposal aims (1) to perform a definitive efficacy study of PSF by comparing 6-month biochemically confirmed abstinence rates in subjects randomized to PSF vs. standard care in a cohort of 450 PLWH smokers, (2) to determine the sociobehavioural moderators and mediators associated with successful cessation, and (3) to complete a careful cost analysis of PSF in order to estimate the incremental cost per quit associated program participation.

If PSF is proven to be effective it will establish a new treatment option for PLWH smokers. Determination of moderators and mediators of program success will provide insight into the mode of action of the intervention and will help guide the development of additional treatment strategies in the future. Finally, the cost analyses will provide critical information about the feasibility of program dissemination and implementation.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infection
* Receives care at Montefiore Medical Center or Georgetown University
* Motivated to quit
* Willing to attend eight 90 minute group sessions

Exclusion Criteria:

* Pregnancy or breastfeeding
* Contraindication to nicotine patch use

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
6 month abstinence from cigarettes | 6 months
  Biochemically-confirmed 7-day point-prevalence abstinence from cigarettes at the 6-month timepoint

SECONDARY OUTCOMES:
Cost per incremental quit | 6 months
  Estimated cost per incremental quit

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Shuter, MD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Montefiore Medical Center, The Bronx, New York

REFERENCES:
- [Background] Moadel AB, Bernstein SL, Mermelstein RJ, Arnsten JH, Dolce EH, Shuter J. A randomized controlled trial of a tailored group smoking cessation intervention for HIV-infected smokers. J Acquir Immune Defic Syndr. 2012 Oct 1;61(2):208-15. doi: 10.1097/QAI.0b013e3182645679. PMID 22732470
- [Derived] Mdege ND, Shah S, Dogar O, Pool ER, Weatherburn P, Siddiqi K, Zyambo C, Livingstone-Banks J. Interventions for tobacco use cessation in people living with HIV. Cochrane Database Syst Rev. 2024 Aug 5;8(8):CD011120. doi: 10.1002/14651858.CD011120.pub3. PMID 39101506

DOCUMENTS (1):
  • Informed Consent Form (2017-01-03): https://cdn.clinicaltrials.gov/large-docs/72/NCT02072772/ICF_000.pdf